CLINICAL TRIAL: NCT02156245
Title: Evaluation of the Effects of Eccentric Training on a Cycle Ergometer, Versus Conventional Concentric Training
Acronym: ENERGETIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CASILLAS DB 2011
Record Dates: First submitted 2014-03-05; First posted 2014-06-05 (Estimated); Last update posted 2019-07-22 (Actual); Status verified 2019-07

CONDITIONS: Readaptation to Effort; Coronaropathy; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "Conventional" group (Experimental)
  Interventions: Other: conventional rehabilitation program (including concentric cycle ergometer)
- "Combined" group (Experimental)
  Interventions: Other: cycling included into a conventional rehabilitation program

INTERVENTIONS:
Other: conventional rehabilitation program (including concentric cycle ergometer)
  Arms: "Conventional" group
Other: cycling included into a conventional rehabilitation program
  Arms: "Combined" group

SUMMARY:
The aim of this study is to assess the efficacy of a rehabilitation protocol based on individualized combined eccentric and concentric cycle ergometer training compared to classical concentric cycle training among patients with either coronary artery disease (CAD) or chronic obstructive pulmonary disease (COPD). This study will therefore evaluate the efficacy of combined eccentric/concentric training on physical capacity and overall autonomy, and will analyse the adaptive mechanisms with regard to both adaptation to cardiac and muscular effort and tolerance.

DETAILED DESCRIPTION:
The research will take place in 3 phases:

PHASE 1 :

30 healthy volunteers will be included to test tolerance to personalized exercise on an eccentric cycle ergometer.

PHASE 2 :

15 patients suffering from coronary artery disease (CAD) and 15 patients suffering from chronic obstructive pulmonary disease (COPD) will be included to test the same protocol.

PHASE 3 :

A total of 169 patients split into 2 parallel groups will be included: a group receiving conventional rehabilitation (group A) and the other group receiving eccentric exercise combined to conventional rehabilitation (group B).

Coronary patients: 93 patients will be included (62 patients in group A and 31 in group B).

COPD patients: 76 patients will be included (38 patients per group).

ELIGIBILITY:
Inclusion Criteria:

* Persons who have provided written informed consent

Healthy volunteers:

* Men or women aged between 40 and 75 years.

Patients with CAD:

* Men or women aged between 40 and 75 years, with coronary artery disease without heart failure referred for a rehabilitation program.
* Left ventricular ejection fraction on echocardiography (Simpson methode) > 45 %

Patients with Chronic obstructive pulmonary disease:

* Men or women aged between 40 and 75 years
* Severe Chronic obstructive pulmonary disease (post-bronchodilatator FEV1/FVC < 0.70 and FEV1 ≤ 60% of predicted value)
* Patient not on oxygen therapy (24h/24)

Exclusion Criteria:

* Person without national health insurance cover
* Severe, obstructive cardiopathy
* Severe aortic valve stenosis,
* Severe progressive heart rhythm or conduction disorders not corrected by a pacemaker and detected during the initial effort test
* Cardiac intracavitary thrombus,
* Severe pulmonary artery hypertension (PAHT systolic >70mmHg),
* Recent history of venous thromboembolism (previous 3 months),
* Impaired executive functions making it impossible to understand and adhere to a rehabilitation program (Mini Mental Test < 24),
* Heart transplant,
* Associated medical condition that could substantially affect functional capacities (examples: non-stabilized metabolic disorders such as progressive renal insufficiency, major asthenia linked to a severe non-stabilized disorder such as neoplasia, systemic disease…).
* Physical incapacity of the lower limbs that could impair rehabilitation, whether they are neurological (central or peripheral), arterial (in particular, peripheral artery disease with a systolic index < 0.6) or orthopedic (degenerative or inflammatory rheumatism).
* Patients who have taken part (within the previous 6 months) or a currently taking part in a rehabilitation program.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2013-09-16 (Actual); Primary Completion 2019-04-03 (Actual); Study Completion 2019-04-03 (Actual)

PRIMARY OUTCOMES:
For patients with CAD: Distance covered during a 6-minute walk test and triceps surae maximal isometric force | Between the initial evaluation (D0) and the final reconditioning evaluation, assessed up to 8 weeks
For COPD patients : Endurance time at 75 % of peak workload achieved on a cycle ergometer during the initial concentric cardiopulmonary exercise test (CPET) | Between the initial evaluation (D0) and the final reconditioning evaluation, assessed up to 8 weeks

SECONDARY OUTCOMES:
For CAD patients: Functional Independence Measure | Between the initial evaluation (D0) and the final reconditioning evaluation, assessed up to 8 weeks
For CAD patients: Timed up and go test | Between the initial evaluation (D0) and the final reconditioning evaluation, assessed up to 8 weeks
For CAD patients: Step test with gas exchange measurement | Between the initial evaluation (D0) and the final reconditioning evaluation, assessed up to 8 weeks
For CAD patients: Distance covered in the 6-minute walk test | Between the initial evaluation (D0) and the final reconditioning evaluation, assessed up to 8 weeks
For CAD patients: peak VO2 and 1st ventilation adaptation threshold | Between the initial evaluation (D0) and the final reconditioning evaluation, assessed up to 8 weeks
For CAD patients: VO2 measurement during the 6 minute walk test | Between the initial evaluation (D0) and the final reconditioning evaluation, assessed up to 8 weeks
For CAD patients: heart rate and systolic blood pressure | Between the initial evaluation (D0) and the final reconditioning evaluation, assessed up to 8 weeks
For CAD patients: cardiac output measured non-invasively | Between the initial evaluation (D0) and the final reconditioning evaluation, assessed up to 8 weeks
For CAD patients: maximum isometric muscle strength of the triceps and quadriceps | Between the initial evaluation (D0) and the final reconditioning evaluation, assessed up to 8 weeks
For CAD patients: tissue oxygenation measured by infrared spectroscopy (non-invasive) at the quadriceps | Between the initial evaluation (D0) and the final reconditioning evaluation, assessed up to 8 weeks
For CAD patients: reaction hyperaemia in the circumflex humeral artery mesured by ultrasound | Between the initial evaluation (D0) and the final reconditioning evaluation, assessed up to 8 weeks
For CAD patients: Measurement of lactates | Between the initial evaluation (D0) and the final reconditioning evaluation, assessed up to 8 weeks
For COPD patients: Distance covered in the 6-minute walk test | Between the initial evaluation (D0) and the final reconditioning evaluation, assessed up to 8 weeks
For COPD patients: peak VO2 and 1st ventilation adaptation threshold | Between the initial evaluation (D0) and the final reconditioning evaluation, assessed up to 8 weeks
For COPD patients: SpO2 and heart rate measurement before, during and after the 6-minute walk test | Between the initial evaluation (D0) and the final reconditioning evaluation, assessed up to 8 weeks
For COPD patients: SpO2 measurement and heart rate during the sessions (warm-up, end of session) | Between the initial evaluation (D0) and the final reconditioning evaluation, assessed up to 8 weeks
For COPD patients: maximum isometric muscle strength of the quadriceps | Between the initial evaluation (D0) and the final reconditioning evaluation, assessed up to 8 weeks
For COPD patients: arterial compliance (pulse wave velocity measurement) | Between the initial evaluation (D0) and the final reconditioning evaluation, assessed up to 8 weeks
For COPD patients: Measurement of lactates | Between the initial evaluation (D0) and the final reconditioning evaluation, assessed up to 8 weeks
For COPD patients: muscle composition and vascularization through muscle biopsies (optional) | Between the initial evaluation (D0) and the final reconditioning evaluation, assessed up to 8 weeks
For COPD patients: St George's Respiratory Questionnaire (SGRQ) | Between the initial evaluation (D0) and the final reconditioning evaluation, assessed up to 8 weeks
For COPD patients: Quality of life-BPCO (VQ11) | Between the initial evaluation (D0) and the final reconditioning evaluation, assessed up to 8 weeks
For COPD patients: COPD Assessment Test (CAT) | Between the initial evaluation (D0) and the final reconditioning evaluation, assessed up to 8 weeks
For COPD patients: BDI/TDI and mMRC dyspnea assessment | Between the initial evaluation (D0) and the final reconditioning evaluation, assessed up to 8 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHU de BESANCON, Besançon
  - CHU de DIJON, Dijon